CLINICAL TRIAL: NCT02645565
Title: Comparison of Intravenous Low Dose Versus High Dose Cyclophosphamide as Induction Therapy in the Treatment of Proliferative Lupus Nephritis
Brief Title: Comparison of Low Dose Versus High Dose Cyclophosphamide as Induction Therapy in the Treatment of Lupus Nephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Dr. Vir Singh Negi, Head of the department and Proffessor of Clinical Immunology, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JIP/IEC/SC/2013/5/435
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Cyclophosphamide; Azathioprine; Methylprednisolone; Prednisolone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose Cyclophosphamide (Active Comparator): Intravenous Cyclophosphamide therapy 500 mg intravenous 2 weekly for 3 months followed by azathioprine 2 mg/kg. Injectable methylprednisolone 1 gm pulse will be given for 3 days before starting the first pulse of cyclophosphamide followed by oral prednisolone 1 mg/kg for 4 weeks and then tapering 5 mg every 2 weeks till 7.5 mg/day.
  Interventions: Drug: Cyclophosphamide; Drug: Azathioprine; Drug: Methylprednisolone
- High Dose Cyclophosphamide (Active Comparator): Intravenous Cyclophosphamide therapy 750mg/m2 intravenous 4 weekly for 6 months followed by azathioprine 2mg/kg. Injectable methylprednisolone 1 gm pulse will be given for 3 days before starting the first pulse of cyclophosphamide followed by oral prednisolone 1 mg/kg for 4 weeks and then tapering 5 mg every 2 weeks till 7.5 mg/day.
  Interventions: Drug: Cyclophosphamide; Drug: Azathioprine; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide is an alkylating agent used for the treatment of lupus nephritis.
  Other Names: Endoxan
Drug: Azathioprine — azathioprine will be given at 2 mg/kg.
  Other Names: Imuran
Drug: Methylprednisolone — Each treatment arm shall receive 1 gm methylprednisolone pulse for 3 days followed by prednisolone 1 mg/kg for 4 weeks and tapered 5 mg every 2 weekly ,to maintain 7.5 mg dose daily
  Other Names: prednisolone,steroid

SUMMARY:
This study will be conducted to find out whether low dose or high dose cyclophosphamide therapy is effective in the treatment of proliferative lupus nephritis.It will also compare the side effects and risks of infection in low dose and high dose cyclophosphamide group. Half of the participants will receive a low dose cyclophosphamide for 3 months and half will receive high dose cyclophosphamide therapy monthly for 6 months followed by azathioprine 2 mg/kg.

DETAILED DESCRIPTION:
The study will be conducted at the Department of Clinical Immunology, Jawaharlal Institute of Postgraduate Medical Education & Research (JIPMER). Once the patients are diagnosed to have systemic lupus erythematosus (SLE) lupus nephritis and they satisfy the inclusion criteria , they will be informed about the nature and severity of the disease and about the expected treatment options and the duration of treatment. After providing written informed consent, eligible patients will be stratified into two groups. Block randomization will be done to generate random allocation sequence.They will receive either a low dose or high dose Cyclophosphamide as per the protocol mentioned below:

Group I : Low dose arm : Intravenous cyclophosphamide fixed pulse 500 mg each 2 weekly total 6 doses followed by azathioprine 2 mg/kg.

Group II : High Dose arm : Intravenous cyclophosphamide therapy 750 mg/m2 will be given every 4 weekly for total 6 doses followed by azathioprine 2 mg/kg.

Intravenous methylprednisolone pulses 1 gm each will be given for 3 days in both the treatment arms followed by prednisolone 1 mg/kg for 4 weeks and then tapering 5 mg every 2 weeks.

Additional drugs as per indication like hydroxychloroquine, antihypertensives and cotrimoxazole prophylaxis shall also be given unless contraindicated.

There will be monitoring of treatment efficacy and side effects in each treatment arm

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of SLE according to the American College of Rheumatology (ACR) criteria
2. Age >16 years
3. Proteinuria ≥500 mg in 24 hours/ urine routine microscopy showing active cellular casts/sediments.
4. Biopsy-proven proliferative lupus glomerulonephritis of class III, IV according to the International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria.

Exclusion Criteria:

1. Patients ever treated previously with intravenous or oral cyclophosphamide or received steroids >15mg/day in the last 3 months.
2. Patients with renal thrombotic microangiopathy, preexisting chronic renal failure, pregnancy, previous malignancy (except skin and cervical intraepithelial neoplasia), diabetes mellitus or coronary heart disease.
3. Patients with previously documented severe toxicity to immunosuppressive drugs.
4. Patients with acute/chronic infections.
5. Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessment of Primary Renal Response | 12 months
  Renal response as by the EULAR guidelines will be evaluated at 12 months for low dose group and high dose cyclophosphamide group. Inactive urinary sediments defined by ≤5 red blood cells (RBC)/hpf, ≤5 white blood cells (WBC)/hpf and no cellular casts as per the American college of rheumatology (ACR) definition.
  1. Complete Response (CR) with urine protein creatinine ratio(UPCR) <0.5 gm and Normal (GFR > 90 ml/min) or stable (<10% deterioration from baseline if GFR was previously abnormal) renal function and inactive urinary sediments.
  2. Partial Response(PR) , defined as ≥50% reduction in proteinuria to subnephrotic levels , normal (GFR > 90 ml/min) or stable (<10% deterioration from baseline if GFR was previously abnormal) renal function and inactive urinary sediments.
  3. No Response : Patients will be classified as non responders if criteria for CR or PR are not met and or if they experience severe flare.

SECONDARY OUTCOMES:
Proportion of patients with Renal and Non renal disease flares | 12 months
  Nephritic flares consist of a reproducible increase in serum creatinine (SCr) concentration of 30% or more (or a reduction in glomerular filtration rate [GFR] by 10% or more) and active urine sediment with an increase in glomerular hematuria by 10 or more red blood cells per high power field, irrespective of changes in UPCR. Proteinuric flares consist of a reproducible doubling of urine protein to creatinine ratio (UPCR) to more than 1.0 after complete renal response or a reproducible doubling of UPCR to more than 2.0 after partial response.
Assessment of adverse events | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Vir Singh Negi, DM, Principal Investigator — Jawaharlal Institute of Postgraduate Medical Education & Research; Dr. Sonal Mehra, MD, Study Chair — Jawaharlal Institute of Postgraduate Medical Education & Research
Locations (1):
- Department of Clinical Immunology , Jawaharlal Institute of Post graduate Medical Educationa and Research, Puducherry, Puducherry, India

REFERENCES:
- [Derived] Mehra S, Usdadiya JB, Jain VK, Misra DP, Negi VS. Comparing the efficacy of low-dose vs high-dose cyclophosphamide regimen as induction therapy in the treatment of proliferative lupus nephritis: a single center study. Rheumatol Int. 2018 Apr;38(4):557-568. doi: 10.1007/s00296-018-3995-3. Epub 2018 Feb 15. PMID 29450636